CLINICAL TRIAL: NCT00228202
Title: Cytomegalovirus Glycoprotein B Genotypes in Israeli Patients: Relationship Between CMV Genotype, Clinical and Demographic Factors
Brief Title: Genotyping of Cytomegalovirus From Patients in Israel
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Other Study IDs: SHEBA-05-3867-NK-CTIL; Sara Orzi MSc thesis
Record Dates: First submitted 2005-09-26; First posted 2005-09-28 (Estimated); Last update posted 2006-08-18 (Estimated); Status verified 2006-01

CONDITIONS: Cytomegalovirus Infections
Keywords: cytomegalovirus; CMV; pregnancy; amniotic fluid; bone marrow; transplantation; viral load; glycoprotein B; genotyping; PCR; real-time PCR; CMV disease; Congenital CMV infection
MeSH Terms: conditions — Cytomegalovirus Infections

STUDY DESIGN:
Observational Model: Natural History | Time Perspective: Other

SUMMARY:
The researchers select 100 cytomegalovirus (CMV) DNA samples from patients diagnosed with CMV infection. Patients include bone marrow transplant patients, pregnant women and newborns. The researchers determine viral load by real-time polymerase chain reaction (PCR). They amplify CMV-gB sequences by PCR and type by sequencing and restriction fragment length polymorphism (RFLP). The researchers obtain clinical data from patients' records. They examine association between patients' clinical status and CMV-gB genotype and viral load.

DETAILED DESCRIPTION:
The study aims at finding association between CMV viral load and viral glycoprotein B genotype and the clinical status of patients suffering from CMV infection. Bone marrow transplant patients are at increased risk of developing severe CMV disease and are routinely followed for viral load. Fetuses are also at high risk for developing severe malformations and neurological defects following maternal primary infection during pregnancy. Therefore amniotic fluid from women diagnosed with CMV infection is examined for CMV presence. Newborns having congenital defects are tested for CMV excretion.

There is not yet any confirmed marker for assessment of the potential severity of the viral infection and for prognosis. Therefore we shall attempt to find association between the viral load and genotype and the clinical status.

CMV DNA samples prepared at the Central Virology Laboratory from clinical specimens obtained from patients for diagnostic purposes will be coded and then subjected to viral load analysis using real-time PCR. The gB genotype will be determined by either of two methods described in the literature: (a) PCR and RFLP (b) PCR and sequencing.

Relevant clinical data will be retrieved from the patients clinical records and saved as coded information to match the samples. Bone marrow transplant patients will be followed for prolonged periods covering repeated viral reactivation events. Clinical records from mothers and newborns will be matched when present. Otherwise maternal and newborn samples will be kept as is.

Statistical analysis will be performed to try and find association between the clinical status of patients, the viral load and the viral genotype.

ELIGIBILITY:
Inclusion Criteria:

* CMV DNA sample from a transplant patient with CMV disease.
* CMV DNA from amniotic fluid of women with CMV infection
* CMV DNA from urine of newborns with congenital defects compatible with CMV.

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100
Dates: Start 2005-09

CONTACTS AND LOCATIONS:
Overall Officials: Naty Keller, MD/PhD, Study Director — Sheba Medical Center
Locations (1):
- Central Virology Laboratory, Chaim Sheba Medical Center Tel-Hashomer, Ramat Gan, Israel